CLINICAL TRIAL: NCT05216653
Title: Preoperative Short-course Radiation Followed by Envafolimab Plus CAPEOX for MSS Locally Advanced Rectal Adenocarcinoma (PRECAM): an Open Label, Prospective, Single Arm Clinical Trial
Brief Title: Preoperative Short-course Radiation Followed by Envafolimab Plus CAPEOX for MSS Locally Advanced Rectal Adenocarcinoma (PRECAM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Vice director, Colorectal Surgery, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220111-8
Record Dates: First submitted 2022-01-14; First posted 2022-01-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: MSS Locally Advanced Rectal Adenocarcinoma
Keywords: Radiation; Envafolimab
MeSH Terms: interventions — envafolimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Short-course Radiation followed by Envafolimab plus CAPEOX (Experimental): The enrolled patients with MSS-type advanced middle-low rectal cancer will receive a combined regimen of neoadjuvant chemoradiotherapy combined with immunotherapy and total mesorectal excision (TME surgery).
  1. Radiotherapy uses a short-range mode, irradiating the primary tumor and high-risk areas with dose of 25 Gy.
  2. After radiotherapy, PD-L1 antibody (150mg/week, subcutaneous injection × 6 weeks) immunotherapy combined with two courses of CAPEOX chemotherapy was performed.
  3. Two weeks after the end of the combined treatment plan in step 2), TME surgery is performed.
  Interventions: Drug: Envafolimab; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Short-course Radiation; Procedure: TME surgery, total mesorectal excision

INTERVENTIONS:
Drug: Envafolimab — This product is administered by subcutaneous injection. The recommended dose of subcutaneous injection is 150 mg, administered weekly (QW).
  Other Names: KN053
Drug: Oxaliplatin — 130mg/m2，ivgtt，d1
Drug: Capecitabine — 1000mg/m2，po，bid，d1-14
Radiation: Short-course Radiation — Short-course radiotherapy, using three-dimensional conformal or intensity-modulated radiotherapy, the dose is divided into 5Gy/f, the total dose is 25Gy/5f, 1f/d, and the irradiation is completed within 7 days.
Procedure: TME surgery, total mesorectal excision — The surgical method can choose open, laparoscopic or robotic according to the specific condition of the patient.

SUMMARY:
Short-course radiotherapy combined with immunotherapy may bring revolutionary changes to the preoperative neoadjuvant treatment mode for locally advanced rectal cancer. According to the existing theory, the use of PD-L1 monoclonal antibody after short-course radiotherapy may be the best solution. In this study, the investigators will perform single-cell sequencing of participants tissue samples, fully explore the multi-dimensional omics information of tumors and microenvironments, explore the characteristics of the treatment benefit population, and try to construct an efficacy prediction model to screen the treatment benefit population early and implement precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to receive neoadjuvant therapy.
2. ≧18 years old.
3. Diagnosed by digital rectal examination, colonoscopy, and high-resolution MRI of the pelvis, the tumor is less than or equal to 12 cm from the anus.
4. Histologically diagnosed as rectal adenocarcinoma.
5. The clinical staging by pelvic contrast-enhanced CT and pelvic high-resolution MRI were cT2-4a N+, cT3/T4a N0.
6. MMR protein detection or MSI gene detection of rectal cancer specimens confirmed pMMR or MSS before treatment .
7. The patient has good compliance and can come to the hospital for re-examination as required.
8. ECOG Scale of Performance Status score 0-1 point.
9. Have not received anti-tumor and immunotherapy before enrollment.
10. Laboratory inspections must meet the following standards:

    1. White blood cell count>3.5×109/L, absolute value of neutrophils>1.8×109/L, platelet count ≥75×109/L, hemoglobin ≥100g/L;
    2. INR≤1.5, and APTT≤1.5 times the upper limit of normal or partial prothrombin time (PT) ≤1.5 times the upper limit of normal;
    3. Total bilirubin ≤ 1.25 times the upper limit of normal; ALT and AST < 5 times the upper limit of normal;
    4. 24h creatinine clearance >50mL/min or serum creatinine <1.5 times the upper limit of normal.
11. Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. History of other malignant diseases in the past 5 years.
2. Patients with metastases from other sites (stage IV patients).
3. Patients with clinical staging of T1-2N0 or T4b, or positive lateral lymph nodes by pelvic contrast-enhanced CT and pelvic high-resolution MRI.
4. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. requiring emergency surgery.
5. Known allergic to oxaliplatin, capecitabine, PD-L1 monoclonal antibody and other drugs.
6. Pathologically suggested signet ring cell carcinoma and mucinous adenocarcinoma.
7. dMMR or MSI-H patients.
8. The patient is accompanied by any unstable systemic disease, including but not limited to: severe infection, uncontrolled diabetes, hypertension uncontrolled by medication, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial Infarction, congestive heart failure, severe cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease; disease affecting the patient's life.
9. The disease (such as mental illness, etc.) or condition (such as alcoholism or drug abuse, etc.) associated with the patient will increase the risk of the patient receiving the trial drug treatment or affect the patient's compliance with the trial requirements, or may confuse the research results.
10. Active autoimmune disease that may worsen while receiving immunostimulants.
11. Known history of positive HIV test or known acquired immunodeficiency syndrome.
12. Patients who are using immunosuppressive agents, except for the following conditions:

    1. Intranasal, inhaled, topical steroids, or topical steroid injections (eg, intra-articular injections);
    2. Physiological doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent;
    3. Steroids used to prevent allergic reactions (eg, before CT scan).
13. Received any other experimental drug treatment or participated in another interventional clinical trial within 30 days before screening
14. Women who are pregnant or breastfeeding or who plan to become pregnant or breastfeeding during the study period; men or women who are unwilling to take effective contraceptive measures.
15. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, etc.
16. Other conditions that the investigator judges that the patient is not suitable to participate in the clinical study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the pathologic complete response (pCR) rate following short-course radiation then Envafolimab Plus CAPEOX | Up to 10 weeks (once surgery is done)
  pCR was defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0).

SECONDARY OUTCOMES:
Tumor regression grade following short-course radiation then Envafolimab Plus CAPEOX as assessed by AJCC/CAP TRG system | Up to 10 weeks (once surgery is done)
  Tumor Regression Grade（TRG）will be done via pathologic assessment on the surgical specimen with AJCC/CAP TRG system
The proportion of participants who remain survival at 3 years | Up to 3 years
  Defined as the percentage of patients alive after 3-year follow-up
The proportion of participants who remain progression free at 3 years | Up to 3 years
  Defined as the percentage of patients without disease recurrence or progression after 3-year follow-up
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | Up to 3 years
  Treatment- related adverse events are assessed by NCI-CTCAE v5.0 in each visit
Surgical Complications of total mesorectal resection procedure for patients after short-course radiation then Envafolimab Plus CAPEOX as assessed by Clavien-Dindo classification | Up to 24 weeks
  Surgical Complications are assessed by Clavien-Dindo classification after surgery.
Quality of life of the patients in a neoadjuvant setting of short-course radiation then Envafolimab Plus CAPEOX as assessed by FACT-C questionnaire | Up to 3 years
  Quality of life is measured via FACT-C questionnaire in each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Dai, MD&PhD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided